CLINICAL TRIAL: NCT05447338
Title: Effectiveness of Post Muscle Inhibition Specific Joint Mobilization on Range of Motion and Pain in Patients With Mechanical Neck Pain
Brief Title: Manual Therapy in Patients With Neck Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional de Córdoba (Other)
Responsible Party: Principal Investigator, Franco Catelotti, Principal Investigator, Universidad Nacional de Córdoba
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 4241
Record Dates: First submitted 2022-05-25; First posted 2022-07-07 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Neck Pain
Keywords: Neck Pain; Rehabilitation; Therapy
MeSH Terms: conditions — Neck Pain | interventions — Nuclear Receptor Subfamily 4, Group A, Member 3

STUDY DESIGN:
Intervention Model Description: The sample will be divided into three intervention groups. Two experimental groups and a control group. Experimental group A: Will receive as treatment the specific joint mobilization technique post muscle inhibition (MAEPI). Experimental group B: Will receive the MAEPI technique as treatment and myofascial induction techniques will be added. The control group: will receive two techniques whose effectiveness is scientifically proven. Which are: Maitland central posterior-anterior passive joint mobilization in C2 + Sustained natural apophyseal sliding (SNAG) in rotation on C1.
Who Masked: Participant
Masking Description: The selection of the intervention group will be made by lottery. The participant will not know to which intervention group they will belong, that is, they will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Specific joint mobilization post muscle inhibition on C1 and C2 (Experimental): Experimental technique alone, with its two variants. That applies a sliding of the articular surfaces of the atlas and axis after a muscular reflex inhibition (proprioceptive neuromuscular facilitation). Between 1 and 5 mobilizations will be carried out per variant of the technique. There will be 4 treatment sessions distributed over 2 weeks.
  Interventions: Procedure: Specific joint mobilization post muscle inhibition on C1; Procedure: Specific joint mobilization post muscle inhibition on C2
- Specific joint mobilization post muscle inhibition on C1 and C2 + myofascial inductions (Experimental): Experimental technique alone, with its two variants. That applies a sliding of the articular surfaces of the atlas and axis after a muscular reflex inhibition (proprioceptive neuromuscular facilitation). Between 1 and 5 mobilizations will be carried out per variant of the technique. Myofascial inductions will also be applied to the cranial and cervical fascia, as well as to the suboccipital, pectoral, angular scapula, sternocleidomastoid, trapezius, internal and external pterygoid, masseter and temporal muscles. There will be 4 treatment sessions distributed over 2 weeks.
  Interventions: Procedure: Specific joint mobilization post muscle inhibition on C1; Procedure: Specific joint mobilization post muscle inhibition on C2; Procedure: Myofascial inductions; Suboccipital induction; Procedure: Myofascial inductions; Synchronization of the temporal bones PHASE 1; Procedure: Myofascial inductions; Horizontal induction of the TMJ.; Procedure: Myofascial inductions; Posterior elongation of the cervical fascia in the supine position; Procedure: Myofascial induction; Angle of the scapula; Procedure: Myofascial induction sternocleidomastoid muscles; Procedure: Myofascial induction of pectoralis major and minor; Procedure: Myofascial induction; upper trapezius; Procedure: Myofascial induction, of the fascia of the subscapularis muscle; Procedure: Intraoral myofascial induction of the masseter; Procedure: Deep myofascial induction of the external pterygoid; Procedure: Intraoral mifascial induction of the internal pterygoid; Procedure: Myofascial inductions; Synchronization of the temporal bones PHASE 2
- Maitland C2 + SNAG C1 (Active Comparator): The Maitland technique will be applied, central postero-anterior passive joint mobilization in the C2 vertebra. As well as the sustained apophyseal slip technique (SNAG) in rotation on C1. The dosage is from 1 to 5 mobilizations per technique. There will be 4 treatment sessions distributed over 2 weeks.
  Interventions: Procedure: Maitland C2; Procedure: SNAG C1

INTERVENTIONS:
Procedure: Specific joint mobilization post muscle inhibition on C1 — Grasp the hand with the thumb or forefinger at the spinous process of C1. The contratoma hand is placed in forceps with the thumb and forefinger on the patient's temple, one on each side. Resisting with the hand on the temple, the therapist asks the patient to perform a 6-second isometric contraction of the cervical spine flexor muscles. The therapist then instructs the patient to relax the musculature and simultaneously performs posteroanterior pressure on the spinous process of C2 and passive extension of the head (with the hand on the temple). The maneuver is repeated until the therapist notices the release in the flexion-extension movement of the head.
  Arms: Specific joint mobilization post muscle inhibition on C1 and C2; Specific joint mobilization post muscle inhibition on C1 and C2 + myofascial inductions
Procedure: Maitland C2 — Maitland central posterior-anterior passive joint mobilization at C2: The patient will lie prone, the therapist behind the patient's head, with both thumbs will apply a central force on the spinous process of C2. The duration of the application will be up to five applications of 10 to 30 seconds in duration, depending on clinical judgment.
  Arms: Maitland C2 + SNAG C1
Procedure: SNAG C1 — Sustained natural apophyseal slippage (SNAG) will be applied e.g. in the case of wanting to improve the left rotation. The therapist performs a sustained anterior glide to the C1 transverse process on the left. The participant will be seated, simultaneously rotating their head to the left while holding the SNAG. The glide of C1 will be maintained by the therapist until the participant's head returns to the neutral starting position. The same will be done, but in the opposite direction to improve the right rotation.
  Arms: Maitland C2 + SNAG C1
Procedure: Specific joint mobilization post muscle inhibition on C2 — The therapist rotates the head to the right side until the final sensation of the movement is noted, either due to pain or muscular tension. From this position, the therapist asks the patient to rotate the head to the left side while offering resistance with both hands in the opposite direction, in such a way as to generate an isometric contraction of the rotator muscles of the head to the left. The therapist then asks the patient to hold the position for 6 seconds. Subsequently, the therapist with the finger in the transverse process of C1, pushes it in the postero-anterior direction and simultaneously (with the contratome hand) rotates the patient's head to the right. The technique is repeated until the ROM improves, always taking into account the patient's tolerance.
  Arms: Specific joint mobilization post muscle inhibition on C1 and C2; Specific joint mobilization post muscle inhibition on C1 and C2 + myofascial inductions
Procedure: Myofascial inductions; Suboccipital induction — The therapist places his hands under the patient's head in such a way that he can palpate the spinous processes of the cervical vertebrae with his fingers. Next, slowly bring your fingers up until they contact the occipital condyles. At this time he should gently move his fingers downward, thus finding the space between the condyles and the spinous process of the axis. Next, flexing the metacarpophalangeal joints to 90°, slowly elevate the skull. The therapist's hands should remain together and the base of the skull should rest on their palms. The therapist should apply pressure with the index, middle and ring fingers of each hand. This pressure should be maintained for a few minutes until a release of the fascia is noted. In the last phase of the technique, the therapist, without releasing the pressure, opens his hands and slowly brings his head back.
  Arms: Specific joint mobilization post muscle inhibition on C1 and C2 + myofascial inductions
Procedure: Myofascial inductions; Synchronization of the temporal bones PHASE 1 — The therapist rests his two forearms on the table, in such a way that he can contact the external auditory canal with his middle fingers. Place the ring fingers on the mastoid processes and the index fingers on the zygomatic arches. Subsequently, a rotary movement is made on the axis marked by the line that joins the middle fingers. With one of the hands, the movement is in the direction of movement clockwise, and with the other hand, simultaneously, in the opposite direction. By obtaining a symmetry in the movement in opposite directions, the movement is made in the same direction with both hands, first forwards and then backwards. Note how the ring fingers rotate first backwards and then upwards. Symmetry in movements should also be sought
  Arms: Specific joint mobilization post muscle inhibition on C1 and C2 + myofascial inductions
Procedure: Myofascial inductions; Horizontal induction of the TMJ. — The therapist places the middle fingers of both hands on the lingual aspect of the lower molar teeth and then gently presses towards the table. This pressure must be maintained for a minimum of 90 to 120 seconds. Afterwards, the therapist, very attentive to the changes in the direction of the fascial restriction, follows the release movement.
  Arms: Specific joint mobilization post muscle inhibition on C1 and C2 + myofascial inductions
Procedure: Myofascial inductions; Posterior elongation of the cervical fascia in the supine position — Position of the patient, lying on the stretcher in the supine position. Therapist position: Sitting at the head of the table. Technique: With one of his hands, the therapist supports the patient's head on the occipital area and slowly brings it to flexo-elevation. With the other hand, he contacts the mass of the paravertebral muscles, placing the thumb on one side of the spine and the proximal interphalangeal joint of the index finger in flexion on the other. While one hand holds the head position, the other performs a downward vertical slide. The maneuver is repeated between 3 and 7 times in a slow and progressive manner.
  Arms: Specific joint mobilization post muscle inhibition on C1 and C2 + myofascial inductions
Procedure: Myofascial induction; Angle of the scapula — Position of the patient, supine position, with the arm resting along the trunk. Position of the therapist, standing or sitting at the head of the table. The therapist places one of his hands under the shoulder blade, embracing the lower angle with the fingertips and bringing it slightly cranially. This maneuver frees access to the superior angle of the scapula, which makes it easier for the index and middle fingers of the other hand to contact the insertion of the angle. More sustained pressure is applied to this point, while the hand placed on the scapula moves in the direction of release.
  Arms: Specific joint mobilization post muscle inhibition on C1 and C2 + myofascial inductions
Procedure: Myofascial induction sternocleidomastoid muscles — Objective, release the myofascial restrictions of the fascia of the SCM muscle. Position of the patient, supine position with the head near the upper edge of the stretcher. Therapist position. sitting at the head of the stretcher. Technique: The therapist, with one hand placed on the occipital region, gently rotates the patient's head. The other hand places it on the mass of the SCM muscle with the thumb at the point of insertion on the mastoid process. While one hand applies the rotational movement and a slight extension of the head, the other performs a transverse slide over the zone of restriction in the SCM muscle. A longitudinal sliding movement of the SCM muscle can be made between the thumb and forefinger of the executing hand.
  Arms: Specific joint mobilization post muscle inhibition on C1 and C2 + myofascial inductions
Procedure: Myofascial induction of pectoralis major and minor — Objective, release the fascia of the pectoralis major and minor muscle. Position of the patient, supine position, with the arm abducted to about 120 degrees. Position of the therapist, standing next to the patient, at head height. Technique: with his cranial hand, the therapist holds the patient's arm, and with the caudal hand, placed in a prone position, contacts the space between pectoralis major and ribs. This contact is made with the fingertips. The pressure should be maintained for about 5 minutes. As the release occurs, both of the therapist's hands must adjust to the direction of the changes. When detecting the restriction in the pectoralis minor, the penetration should be deepened with the hand, sliding it over the ribs. Contact and restraints with the pectoralis minor and major are often particularly painful, forcing the therapist to apply controlled force.
  Arms: Specific joint mobilization post muscle inhibition on C1 and C2 + myofascial inductions
Procedure: Myofascial induction; upper trapezius — Objective, release the myofascial restrictions of the upper trapezius. Position of the patient, supine, with the elbow flexed and the hand resting on the abdomen, and the arm in a slight abduction. Therapist position, sitting at the head of the table. Technique: The therapist places his hand on the patient's shoulder so that he can grasp the fibers of the upper trapezius between the index, middle, and ring fingers above and the thumb below. Subsequently, he exerts gentle and sustained pressure overcoming three restraining barriers.
  Arms: Specific joint mobilization post muscle inhibition on C1 and C2 + myofascial inductions
Procedure: Myofascial induction, of the fascia of the subscapularis muscle — Position of the patient, supine, with the arm raised about 90-160 degrees, depending on the degree of movement restriction. Therapist position, standing at the head of the table. Phase A With his cranial hand, the therapist holds the patient's arm and performs very gentle traction. The palm of the caudal hand, thumb up, is placed on the outer edge of the scapula, as close as possible to the glenohumeral joint. A slight traction is performed with both hands in opposite directions, subsequently following the direction of release. Phase B, The thumb of the caudal hand slightly invades the space between the inner aspect of the scapula and the thorax. The rest of the application is performed as in phase A. Phase C, the therapist places his caudal hand in a prone position and slowly penetrates the aforementioned space with the tips of the fingers. sustained for a time ranging between 90 seconds and 5 minutes, following the release stages.
  Arms: Specific joint mobilization post muscle inhibition on C1 and C2 + myofascial inductions
Procedure: Intraoral myofascial induction of the masseter — Position of the patient, supine position, on the stretcher without the pillow. Position of the therapist, sitting at the head of the table. Technique: The therapist, with the index of his hand, contacts the masseter just below the zygomatic arch and inside the mouth. To ensure proper contact on the masseter, the patient is asked to attempt to close the mouth. Once the muscle is correctly located, the patient should immediately relax the masseter. Next, the therapist compresses the masseter between his index finger and thumb. You have to wait long enough for the release to occur. Sometimes both hands are used by placing the forefinger of the other hand on the outer surface.
  Arms: Specific joint mobilization post muscle inhibition on C1 and C2 + myofascial inductions
Procedure: Deep myofascial induction of the external pterygoid — Objective, release the myofascial restrictions and recover the functional coordination of the external pterygoid muscles.
  Position of the patient, supine position, on the stretcher without the pillow. Therapist position, sitting at the head of the table. Technique: The therapist palpates the temporomandibular joint with the index or middle finger of one hand. With the index finger of the other hand, he contacts the pterygoid inside the mouth and maintains pressure until release occurs.
  Arms: Specific joint mobilization post muscle inhibition on C1 and C2 + myofascial inductions
Procedure: Intraoral mifascial induction of the internal pterygoid — Objective, release the restrictions of the internal pterygoid fascia. Position of the patient, supine position on the stretcher. Therapist position, sitting laterally at the head of the stretcher and looking at the patient. Technique: Therapist palpates the TMJ with the index or middle finger of one hand. With the index of the other hand, he contacts the pterygoid inside the mouth and maintains pressure until release occurs. You have to wait three consecutive releases.
  Arms: Specific joint mobilization post muscle inhibition on C1 and C2 + myofascial inductions
Procedure: Myofascial inductions; Synchronization of the temporal bones PHASE 2 — The therapist rests his two forearms on the table, in such a way that he can contact the external auditory canal with his middle fingers. Place the ring fingers on the mastoid processes and the index fingers on the zygomatic arches. Subsequently, a rotary movement is made on the axis marked by the line that joins the middle fingers. With one of the hands, the movement is in the direction of movement clockwise, and with the other hand, simultaneously, in the opposite direction. By obtaining a symmetry in the movement in opposite directions, the movement is made in the same direction with both hands, first forwards and then backwards. Note how the ring fingers rotate first backwards and then upwards. Symmetry in movements should also be sought.
  Arms: Specific joint mobilization post muscle inhibition on C1 and C2 + myofascial inductions

SUMMARY:
Neck pain is a common clinical condition of some diseases that affect the soft tissues, musculotendinous structures and joints of the cervical spine. It is characterized by pain in the posterior and lateral muscles of the neck, muscle contractures and partial functional impotence. An important finding is that approximately 60% of total cervical rotation takes place at C1-C2, regardless of age. The test used to diagnose dysfunction of the upper cervical spine is the Cervical Rotation Flexion Test (CRFT) and is measured in degrees through various instruments, the most current validated by scientific literature are mobile applications (Clinometer and Compass ). Having in clear the importance of the location (C1-C2) of the origin of many of the symptoms and signs that cervicalgia generates and mainly the restriction of the range of movement that they produce in the cervical spine. It is that the manual therapy technique: Joint mobilization post muscular inhibition (MAEPI) that is included in this study for its analysis, is directed to this segment of the cervical spine. This differs from other similar techniques, in terms of location and movement of the joint surfaces, which have been previously studied and have shown their effectiveness (techniques that will be used in the control group), in that the micro movements of the joint surfaces ( joint arthrokinematics) based on the principles of Kaltenborn-Evjenth will be combined with the principles of the hold relax technique belonging to the Proprioceptive Neuromuscular Facilitation method. The main therapeutic objective of the MAEPI technique is to improve mobility and reduce pain in the cervical spine.

Hypothesis: The MAEPI technique will improve mobility and reduce neck pain as well as other symptoms associated with neck pain, such as headache, dizziness and nausea, and will be more effective than those of the control group (Maitland central posterior-anterior passive joint mobilization in C2 and natural apophyseal slippage sustained (SNAG) in rotation about Mulligan's C1). The MAEPI technique will be more effective when applied later to myofascial induction techniques.

DETAILED DESCRIPTION:
Main goal

-Determine the effectiveness of the MAEPI applied on C1-C2 on the improvement of the range of motion and pain in patients with mechanical neck pain. As well as its effectiveness after performing myofascial induction techniques.

Specific objectives

* Identify the disability index, the intensity of the pain and the degree of mobility of the patients before and after the application of the proposed treatment protocols.
* Identify other symptoms associated with neck pain, such as dizziness, headache and nausea before and after the application of treatment protocols.
* Establish whether there are significant differences in terms of ROM between the proposed protocols, taking into account age, sex, work activity of individuals with neck pain in relation to evolution.

Sample size: The sample size estimate was based on data from previous studies. The standard deviation of 11.1º of the range of motion of the average of the CRFT measurements in patients with upper cervical dysfunction was used. The calculation was performed using the GRANMO sample size calculator (version 7). For an analysis of variance, accepting an alpha risk of 0.05 and a beta risk of less than 0.2 in a unilateral contrast, 38 subjects are needed in each group to detect a minimum difference of 8º between two groups, assuming that there are 3 groups and a deviation 11.1º standard. A rate of loss to follow-up of 10% has been estimated. In the case of repeated paired means by group (experimental group A, MAEPI), accepting an alpha risk of 0.05 and a beta risk of 0.2 in a bilateral contrast, 16 subjects are required to detect a difference equal to or greater than 8 degrees. A standard deviation of 11.1 is assumed. A rate of loss to follow-up of 0% has been estimated.

Data analysis: The InfoStat program will be used. The data will be analyzed according to the nature of each variable in the ANAVA study, non-linear regression, categorical, correlational data and multiple comparisons test (Fisher's test), establishing significant differences when p<0.05 for all cases. The variables dizziness, headache and nausea: they will be evaluated using a qualitative table and later they will be compared using the Chi square test. In the experimental group A: MAEPI, the t test will be performed for paired data (before and after, for the intervention group of the technique alone).

Expected results

Regarding therapeutic effects, it is expected that:

1. Experimental Group A is superior to the Control Group.
2. Experimental Group B is superior to Experimental Group A.

ELIGIBILITY:
Inclusion criteria:

* You must have a medical indication for cervical physiotherapy.
* Must present decreased ROM of the upper cervical spine assessed with CRFT, either acute or subacute and of a mechanical type or PN and grade I and II of severity according to The Neck Pain Task Force.

Exclusion criteria:

* Joint instability, dislocations, fractures or stenosis of the cervical spinal canal.
* Malformations and/or bony alterations of the cervical spine or the brain.
* Head injury or whiplash in the last 10 years. Infections, unhealed wounds, tumors, vascular pathology or cancer that compromises the cervical spine and/or the brain.
* Being under treatment with anti-inflammatories, muscle relaxants or some type of pain reliever.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 114 (Estimated)
Dates: Start 2021-08-30 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Degrees of movement | After the 6 treatment sessions that will be carried out in a period of two weeks for all groups (week 3)
  The cervical flexion-rotation test (CFRT) will be measured in degrees of motion. CFRT is effective in evaluating the presence/absence of upper cervical spine dysfunction. If there are symptoms and the range is decreased by more than 10º (normal is 44º on each side), the test is considered positive and, therefore, there is a limitation in the C1-C2 level. The instrument that will be used to measure the rotation of the upper cervical spine in degrees will be the Compass mobile application that has been validated to measure cervical ROM. The goal is to measure the change in range of motion before and after treatment.

SECONDARY OUTCOMES:
Neck Disability Index | After the 6 treatment sessions that will be carried out in a period of two weeks for all groups (week 3)
  It is a 10-item questionnaire that measures disability related to a patient's neck pain. Each question is measured on a scale of 0 (no disability) to 5, and an overall score of 100 is calculated by adding the score for each item and multiplying it by two. A higher NDI score means greater patient perceived disability due to neck pain. The "minimum clinically important change" by patients has been found to be 5-10%. The objective is to measure the change in the disability index before and after treatment.

OTHER OUTCOMES:
Numeric pain scale | After the 6 treatment sessions that will be carried out in a period of two weeks for all groups (week 3)
  Numbered scale from 0-10, where 0 is the absence and 10 the greatest intensity; the patient selects the number that best evaluates the intensity of the symptom. It is the simplest and the most used. Numbering Interpretation: 0 = no pain 10 = maximum pain. The objective is to measure the change in pain intensity before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Franco Catelotti, Principal Investigator — Universidad Nacional de Córdoba; Argentina
Locations (1):
- Conci Carpinella, Córdoba, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hall TM, Briffa K, Hopper D, Robinson K. Comparative analysis and diagnostic accuracy of the cervical flexion-rotation test. J Headache Pain. 2010 Oct;11(5):391-7. doi: 10.1007/s10194-010-0222-3. Epub 2010 May 28. PMID 20508964